CLINICAL TRIAL: NCT04974749
Title: An Open-label Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of REPLAGAL® in Treatment-naïve Chinese Subjects With Fabry Disease
Brief Title: A Study of REPLAGAL® in Treatment-naive Chinese Participants With Fabry Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-675-3001; 2022-004246-35 (EudraCT Number)
Record Dates: First submitted 2021-07-21; First posted 2021-07-23 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-07

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- REPLAGAL (Experimental): Participants received REPLAGAL 0.2 milligrams per kilogram (mg/kg) body weight, intravenous (IV) infusion, every other week (EOW) from Day 1 (Week 0) up to Week 52.
  Interventions: Biological: REPLAGAL

INTERVENTIONS:
Biological: REPLAGAL — REPLAGAL IV infusion.
  Other Names: Agalsidase Alfa; TAK-675

SUMMARY:
The main aim of the study is to assess the safety of REPLAGAL. Study participants will receive REPLAGAL as an intravenous infusion every other week for 52 weeks. Participants will visit their study clinic many times throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant and/or legally authorized representative must voluntarily sign an Institutional Review Board/Independent Ethics Committee approved written informed consent form (ICF) after all relevant aspects of the study have been explained and discussed with the participant. For the participants less than (<) 18 years old, participants will give assent AND their parent(s)/legally authorized representative should sign the ICF accordingly.
* The participant has confirmed diagnosis of Fabry disease as determined by the investigator, according to medical record including:

  * For male participant, Fabry disease is confirmed by a deficiency of α-galactosidase A (GLA) activity and a mutation in the GLA gene
  * For female participant, Fabry disease is confirmed by a mutation in the GLA gene.
* The participant is 7 to 65 years of age, inclusive, at screening.
* Female participants of childbearing potential must have a negative pregnancy test at screening.
* Female participants of childbearing potential must agree to use a medically acceptable method of contraception at all times during the study and for at least 14 days after the final investigational product infusion.
* The participant is deemed, as determined by the investigator, to have adequate general health to undergo the specified protocol-related procedures and to have no safety or medical contraindications for participation.
* The participant has not received any treatment (approved or investigational) specific to Fabry disease, such as ERT, chaperone therapy, or substrate reduction therapy.
* The adult participant (greater than or equal to [>=] 18 years old) must have an estimated glomerular filtration rate (eGFR) of 45 to 120 milliliter per minute per 1.73 meter square (mL/min/1.73 m^2) (inclusive). Serum creatinine is tested and the eGFR is calculated by central laboratory using the Chronic Kidney Disease Epidemiology (CKD-EPI) equation.

Exclusion Criteria:

* In the opinion of the investigator, the participant's life expectancy is less than or equal to (<=) 5 years.
* The participant has undergone or is scheduled to undergo kidney transplantation or is currently on dialysis or has any signs or symptoms of end stage renal disease.
* The participant has a urine protein/creatinine ratio of greater than (>) 500 milligram per gram (mg/g).
* The participant has a clinically relevant history of allergy or signs or symptoms of severe hypersensitivity, which in the investigator's judgment, will substantially increase the participant's risk if he or she participates in the study.
* In the opinion of the investigator, the participant has non-Fabry disease-related cause of end organ (renal, cardiovascular, central nervous system) dysfunction/failure or is receiving medications that may affect the rate of disease progression, as assessed by renal measures.
* The participant has a positive test result at screening for hepatitis B surface antigen with detectable hepatitis B viral deoxyribonucleic acid (DNA) load, hepatitis C virus (HCV) antibody with confirmation by HCV ribonucleic acid polymerase chain reaction testing, or human immunodeficiency virus antibody.
* The participant has received prior treatment with any of the following medications, with the exception of non-systemic use:

  * Chloroquine
  * Amiodarone
  * Monobenzone
  * Gentamicin
* The participant is pregnant or lactating.
* The participant has a body mass index >35 kilogram per square meter (kg/m^2).
* The participant is treated or has been treated with any investigational drug for indication other than Fabry disease within 30 days of study start.
* The participant and/or the participant's parent(s)/legal guardian is unable to understand the nature, scope, and possible consequences of the study.
* The participant is unable to comply with the protocol, example, uncooperative with protocol schedule, refusal to agree to all of the study procedures, inability to return for evaluations, or is otherwise unlikely to complete the study, as determined by the investigator.

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (6):
- China (6):
  - Peking Union Medical College Hospital, Beijing
  - Xiangya Hospital, Central South University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - The Children's Hospital of Zhejiang University School of Medicine, Hangzhou
  - Shandong Provincial Hospital, Jinan
  - Ruijin Hospital, Shanghai Jiaotong Uni. School of Med., Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/61031f84beb21d002a926063

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 6 investigative sites in China from 1 May 2022 to 3 January 2024.
Pre-assignment Details: A total of 20 participants with Fabry disease were enrolled in this study to receive REPLAGAL for 52 weeks.
Period: Overall Study
Arm/Group | REPLAGAL
Started | 20
Completed | 17
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Gestation | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Set included all participants who signed the informed consent, were enrolled in the study, and received at least 1 study drug infusion (full or partial).
Groups:
- REPLAGAL: Participants received REPLAGAL 0.2 mg/kg body weight, IV infusion, EOW from Day 1 (Week 0) up to Week 52.
Arm/Group | REPLAGAL
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.1 (14.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 20
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 160.47 (9.271)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 53.88 (10.370)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter square (kg/m^2)] — BMI = weight (kg)/[height (m)^2]
  kilograms per meter square (kg/m^2) | 20.87 (3.674)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that did not necessarily have a causal relationship with this investigational product (IP) or medicinal product. Serious AE was any untoward medical occurrence (whether considered to be related to investigational product or not) that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital abnormality/birth defect, and was an important medical event. A TEAE was defined as any event emerging at or after the initiation of treatment with an IP or any existing event that worsened in either intensity or frequency following exposure to the IP until the end of the safety follow-up period.
Time Frame: From start of study drug administration up to 14 days after end of treatment (EOT) [up to Week 54]
Population: Safety Analysis Set included all participants in the ITT Set who received at least 1 dose of REPLAGAL.
Measure: Count of Participants; unit: Participants
Arm/Group | REPLAGAL
Number analyzed (Participants) | 20
Participants | 2

2. Secondary Outcome: Number of Participants With TEAEs
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that did not necessarily have a causal relationship with this investigational product or medicinal product. A TEAE was defined as any event emerging at or after the initiation of treatment with an IP or any existing event that worsened in either intensity or frequency following exposure to the IP until the end of the safety follow-up period.
Time Frame: From start of study drug administration up to 14 days after EOT (up to Week 54)
Population: Safety Analysis Set included all participants in the ITT Set who received at least 1 dose of REPLAGAL.
Measure: Count of Participants; unit: Participants
Arm/Group | REPLAGAL
Number analyzed (Participants) | 20
Participants | 20

3. Secondary Outcome: Number of Participants With Infusion-related Reactions (IRRs)
Description: An IRR was defined as an event that began either during or within 24 hours after the start of the infusion, and was judged as related to treatment with the IP. An IRR could be serious or non-serious. Adverse events that were considered IRRs were noted as such in the participant's source documentation. Other AEs which occurred prior to the infusion, along with AEs associated with protocol-defined testing and assessments (example, laboratory testing and physical examinations), which were performed prior to the infusion, were not considered as IRRs.
Time Frame: From start of study drug administration up to Week 52
Population: Safety Analysis Set included all participants in the ITT Set who received at least 1 dose of REPLAGAL.
Measure: Count of Participants; unit: Participants
Arm/Group | REPLAGAL
Number analyzed (Participants) | 20
Participants | 5

4. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADA) to REPLAGAL
Description: Number of participants with positive ADA to REPLAGAL were reported.
Time Frame: Baseline up to Week 52
Population: Safety Analysis Set included all participants in the ITT Set who received at least 1 dose of REPLAGAL.
Measure: Count of Participants; unit: Participants
Arm/Group | REPLAGAL
Number analyzed (Participants) | 20
Participants | 6

5. Secondary Outcome: Number of Participants With Positive Neutralizing Antibodies (NAb) to REPLAGAL
Description: Number of participants with positive NAb to REPLAGAL were reported.
Time Frame: Baseline up to Week 52
Population: Safety Analysis Set included all participants in the ITT Set who received at least 1 dose of REPLAGAL.
Measure: Count of Participants; unit: Participants
Arm/Group | REPLAGAL
Number analyzed (Participants) | 20
Participants | 5

6. Secondary Outcome: Number of Participants With Clinically Meaningful Changes in Laboratory Parameters
Description: Laboratory assessment included parameters of serum chemistry, hematology, and urinalysis. Clinically meaningful laboratory parameters assessment was based on investigator interpretation. Number of participants with clinically meaningful changes in laboratory parameters were reported.
Time Frame: From start of study drug administration up to Week 52
Population: Safety Analysis Set included all participants in the ITT Set who received at least 1 dose of REPLAGAL.
Measure: Count of Participants; unit: Participants
Arm/Group | REPLAGAL
Number analyzed (Participants) | 20
Participants | 0

7. Secondary Outcome: Number of Participants With Clinically Meaningful Changes in Vital Signs
Description: Vital sign assessment included pulse, blood pressure, respiratory rate, and temperature. Clinically meaningful vital signs assessment was based on investigator interpretation. Number of participants with clinically meaningful abnormalities in vital signs were reported.
Time Frame: From start of study drug administration up to Week 52
Population: Safety Analysis Set included all participants in the ITT Set who received at least 1 dose of REPLAGAL.
Measure: Count of Participants; unit: Participants
Arm/Group | REPLAGAL
Number analyzed (Participants) | 20
Participants | 0

8. Secondary Outcome: Number of Participants With Clinically Meaningful Changes in Electrocardiogram (ECG) Parameters
Description: ECG parameters included assessment of heart rate, sinus rhythm, atrial or ventricular hypertrophy, and assessment of PR, QRS, QT, and corrected QT intervals. Clinically meaningful ECG assessment was based on investigator interpretation. Number of participants with clinically meaningful abnormalities in 12-lead ECG were reported.
Time Frame: From start of study drug administration up to Week 52
Population: Safety Analysis Set included all participants in the ITT Set who received at least 1 dose of REPLAGAL.
Measure: Count of Participants; unit: Participants
Arm/Group | REPLAGAL
Number analyzed (Participants) | 20
Participants | 0

9. Secondary Outcome: Renal Function as Assessed by Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 52
Description: Renal function was assessed by eGFR using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula for ≥18 years participants, eGFR = 141 x min (Scr/κ,1)^(α) x max(Scr/κ,1)^(-1.209) x 0.993^(Age) x 1.018 (if female) x 1.159 (if black) where: Scr is serum creatinine (milligram per deciliter [mg/dL]); κ is 0.7 for females and 0.9 for males; α is -0.329 for females and -0.411 for males; min indicates the minimum of Scr/κ or 1; max indicates the maximum of Scr /κ or 1. For <18 years participants, Counahan-Barratt equation was used for calculation of eGFR. eGFR = (0.43 × height in centimeter [cm])/Scr where, Scr is serum creatinine (mg/dL). Renal function as assessed by eGFR was expressed using the unit: milliliters/minute/1.73 meter square (mL/min/1.73m^2).
Time Frame: Baseline, Week 52
Population: Modified Intent-to-treat (mITT) Set included all enrolled participants who had received at least 1 dose of investigational product and completed at least 1 post-baseline efficacy assessment of the endpoints.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | REPLAGAL
Number analyzed (Participants) | 19
mL/min/1.73m^2 | 4.1 (12.48)

10. Secondary Outcome: Change From Baseline in eGFR Values at Weeks 8, 16, 28, and 40
Description: The eGFR was calculated by CKD-EPI formula for ≥18 years participants, eGFR = 141 x min (Scr/κ,1)^(α) x max(Scr/κ,1)^(-1.209) x 0.993^(Age) x 1.018 (if female) x 1.159 (if black) where: Scr is serum creatinine (mg/dL); κ is 0.7 for females and 0.9 for males; α is -0.329 for females and -0.411 for males; min indicates the minimum of Scr/κ or 1; max indicates the maximum of Scr /κ or 1. For <18 years participants, Counahan-Barratt equation was used for calculation of eGFR. eGFR = (0.43 × height in cm)/Scr where, Scr is serum creatinine (mg/dL).
Time Frame: Baseline, Weeks 8, 16, 28, and 40
Population: mITT Set included all enrolled participants who had received at least 1 dose of investigational product and completed at least 1 post-baseline efficacy assessment of the endpoints. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | REPLAGAL
Number analyzed (Participants) | 19
mL/min/1.73m^2
  Week 8: number analyzed (Participants) | 18
  Week 8 | -1.2 (15.66)
  Week 16: number analyzed (Participants) | 18
  Week 16 | -0.4 (13.67)
  Week 28: number analyzed (Participants) | 17
  Week 28 | 5.1 (11.25)
  Week 40: number analyzed (Participants) | 16
  Week 40 | 0.3 (13.17)

11. Secondary Outcome: Change From Baseline in Left Ventricular Mass Index (LVMI) at Weeks 16 and 52
Description: LVMI was measured by echocardiography at the clinical sites, and LVMI was derived using the following formula:
  LVM [grams] = 0.8×[1.04×{(LVDd + IVSTd + PWTd)^3 - LVDd^3}] + 0.6, where: LVDd is left ventricular internal diameter (diastolic) (cm), IVSTd is intraventricular septum thickness (diastolic) (cm), and PWTd is posterior wall thickness (diastolic) (cm). LVM indexed to height (LVMI) = LVM/height^2.7 (g/m^2.7), where height was measured in meter.
Time Frame: Baseline, Weeks 16 and 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: grams per meter (g/m)^2.7
Arm/Group | REPLAGAL
Number analyzed (Participants) | 19
grams per meter (g/m)^2.7
  Week 16: number analyzed (Participants) | 14
  Week 16 | -0.4696 (6.81928)
  Week 52: number analyzed (Participants) | 12
  Week 52 | -1.7261 (9.87836)

12. Secondary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF) at Weeks 16 and 52
Description: LVEF is the central measure of left ventricular systolic function. LVEF is the fraction of chamber volume ejected in systole (stroke volume) in relation to the volume of the blood in the ventricle at the end of diastole (end-diastolic volume). This was measured by echocardiography at the clinical sites.
Time Frame: Baseline, Weeks 16 and 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percent of LVEF
Arm/Group | REPLAGAL
Number analyzed (Participants) | 19
percent of LVEF
  Week 16: number analyzed (Participants) | 14
  Week 16 | -1.1 (7.29)
  Week 52: number analyzed (Participants) | 12
  Week 52 | 0.8 (3.28)

13. Secondary Outcome: Change From Baseline in Urine Protein/Creatinine Ratio
Description: The change from baseline in urine protein/creatinine ratio was derived from early morning spot urine samples collected at the specified time points.
Time Frame: Baseline, Weeks 8, 16, 28, 40, and 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: gram per gram
Arm/Group | REPLAGAL
Number analyzed (Participants) | 19
gram per gram
  Week 8: number analyzed (Participants) | 18
  Week 8 | 0.0759 (0.17486)
  Week 16: number analyzed (Participants) | 18
  Week 16 | 0.1061 (0.21743)
  Week 28: number analyzed (Participants) | 16
  Week 28 | 0.0711 (0.16049)
  Week 40: number analyzed (Participants) | 14
  Week 40 | 0.0830 (0.16333)
  Week 52: number analyzed (Participants) | 17
  Week 52 | 0.0627 (0.16508)

14. Secondary Outcome: Change From Baseline in Brief Pain Inventory (BPI) Short Form Pain Severity Total Score
Description: The BPI short form is a numeric rating scale that assesses the severity of pain (severity scale), its impact on daily functioning (Pain Interference scale). BPI short form pain severity scale has been reported here. Pain severity scale has 4 questions that assess pain intensity (worst, least, average, right now) on 10-point rating scales (0=No pain to 10=Pain as bad as you can imagine). The pain severity score is calculated as the average of questions, with a total score ranging from 0 to 10 with higher scores indicating more pain. A negative change from baseline indicates better outcome.
Time Frame: Baseline, Weeks 8, 16, 28, 40, and 52
Population: mITT Set included all enrolled participants who had received at least 1 dose of investigational product and completed at least 1 post-baseline efficacy assessment of the endpoints. Overall number analyzed is the number of participants with pain at baseline. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REPLAGAL
Number analyzed (Participants) | 7
score on a scale
  Week 8 | -1.607 (2.8572)
  Week 16 | -2.214 (2.4041)
  Week 28: number analyzed (Participants) | 6
  Week 28 | -1.833 (2.6957)
  Week 40: number analyzed (Participants) | 6
  Week 40 | -1.375 (2.8007)
  Week 52: number analyzed (Participants) | 6
  Week 52 | -0.958 (3.3370)

15. Secondary Outcome: Change From Baseline in BPI Short Form Pain Interference Total Score
Description: The BPI short form is a numeric rating scale that assesses the severity of pain (severity scale), its impact on daily functioning (Pain Interference scale). BPI short form pain interference scale has been reported here. Pain interference scale has 7 questions that assess impact of pain on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life) on 10-point rating scales as (0=Does not interfere to 10=Completely interferes). The pain interference score is calculated as the average of questions, with a total score ranging from 0 to 10 with higher scores indicating more interference. A negative change from baseline indicates better outcome.
Time Frame: Baseline, Weeks 8, 16, 28, 40, and 52
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REPLAGAL
Number analyzed (Participants) | 7
score on a scale
  Week 8 | -2.286 (3.6636)
  Week 16 | -3.571 (3.9812)
  Week 28: number analyzed (Participants) | 6
  Week 28 | -4.738 (4.3221)
  Week 40: number analyzed (Participants) | 6
  Week 40 | -3.810 (3.8222)
  Week 52: number analyzed (Participants) | 6
  Week 52 | -3.643 (5.7020)

16. Secondary Outcome: Percent Change From Baseline in Plasma Globotriaosylsphingosine (Lyso-Gb3) Level
Description: Plasma lyso-Gb3 determinations were performed at the central laboratory using a validated liquid chromatography-tandem mass spectrometry bioanalytical assay.
Time Frame: Baseline, Weeks 8, 16, 28, 40, and 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | REPLAGAL
Number analyzed (Participants) | 19
percent change
  Week 8: number analyzed (Participants) | 18
  Week 8 | -36.236 (24.7056)
  Week 16: number analyzed (Participants) | 18
  Week 16 | -38.147 (24.7376)
  Week 28: number analyzed (Participants) | 17
  Week 28 | -37.764 (25.8314)
  Week 40: number analyzed (Participants) | 17
  Week 40 | -35.565 (27.7874)
  Week 52: number analyzed (Participants) | 17
  Week 52 | -37.072 (27.5659)

17. Secondary Outcome: Number of Participants With Hearing Loss as Assessed by Audiology Testing
Description: Hearing loss was assessed in participants with the age <18 years old by audiology testing. Audiology testing included pure tone conduction and bone conduction for each ear using 4 different pure tone frequencies (500 hertz [Hz], 1000 Hz, 2000 Hz, and 4000 Hz). Any changes in threshold were to be categorized as conductive, sensorineural, or unknown.
Time Frame: Baseline up to Week 52
Population: mITT Set included all enrolled participants who had received at least 1 dose of investigational product and completed at least 1 post-baseline efficacy assessment of the endpoints. Overall number analyzed is the number of participants with age <18 years old.
Measure: Count of Participants; unit: Participants
Arm/Group | REPLAGAL
Number analyzed (Participants) | 6
Participants | 0

18. Secondary Outcome: Area Under Serum Concentration-time Curve From the Time of Dosing to the Last Measurable Concentration (AUC0-last) of REPLAGAL
Time Frame: Pre-infusion (0 minutes), during infusion (20 minutes) and end of infusion (40 minutes), and post-infusion at 50, 60, 90, 120, 240, and 360 minutes at Weeks 0 and 28
Population: Intensive Pharmacokinetic (PK) Set included participants in the PK Set who provided intensive sampling.
Measure: Mean (Standard Deviation); unit: minutes*units per milliliter (min*U/mL)
Arm/Group | REPLAGAL
Number analyzed (Participants) | 10
minutes*units per milliliter (min*U/mL)
  Week 0 | 229000 (48768)
  Week 28 | 297300 (139640)

19. Secondary Outcome: Area Under Serum Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of REPLAGAL
Time Frame: as for outcome 18
Population: Intensive PK Set included participants in the PK Set who provided intensive sampling.
Measure: Mean (Standard Deviation); unit: min*U/mL
Arm/Group | REPLAGAL
Number analyzed (Participants) | 10
min*U/mL
  Week 0 | 233700 (49553)
  Week 28 | 309500 (157460)

20. Secondary Outcome: Serum Clearance of Administered Dose (CL) of REPLAGAL
Description: Clearance is defined as a quantitative measure of the rate at which a drug substance is removed from the body. CL = dose/AUC.
Time Frame: as for outcome 18
Population: Intensive PK Set included participants in the PK Set who provided intensive sampling.
Measure: Mean (Standard Deviation); unit: milliliters per minute (mL/min)
Arm/Group | REPLAGAL
Number analyzed (Participants) | 10
milliliters per minute (mL/min)
  Week 0 | 187.4 (35.770)
  Week 28 | 195.5 (226.52)

21. Secondary Outcome: Serum Clearance of Administered Dose Normalized Based on Body Weight of REPLAGAL
Description: Clearance is defined as a quantitative measure of the rate at which a drug substance is removed from the body. CL normalized for body weight was reported. CL= (dose/AUC)/ body weight. Clearance was expressed using the unit: milliliters/minute/kilogram (mL/min/kg).
Time Frame: as for outcome 18
Population: Intensive PK Set included participants in the PK Set who provided intensive sampling.
Measure: Mean (Standard Deviation); unit: mL/min/kg
Arm/Group | REPLAGAL
Number analyzed (Participants) | 10
mL/min/kg
  Week 0 | 3.234 (0.78070)
  Week 28 | 3.183 (3.5632)

22. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of REPLAGAL
Time Frame: as for outcome 18
Population: Intensive PK Set included participants in the PK Set who provided intensive sampling.
Measure: Mean (Standard Deviation); unit: units per milliliter (U/mL)
Arm/Group | REPLAGAL
Number analyzed (Participants) | 10
units per milliliter (U/mL)
  Week 0 | 4620.55 (1046.889)
  Week 28 | 4507.99 (1682.041)

23. Secondary Outcome: Terminal Elimination Half-life (T1/2z) of REPLAGAL
Description: T1/2 is defined as the natural log of 2 divided by the terminal rate constant (ƛz).
Time Frame: as for outcome 18
Population: Intensive PK Set included participants in the PK Set who provided intensive sampling.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | REPLAGAL
Number analyzed (Participants) | 10
minutes
  Week 0 | 45.36 (23.058)
  Week 28 | 66.34 (27.272)

24. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) of REPLAGAL
Time Frame: as for outcome 18
Population: Intensive PK Set included participants in the PK Set who provided intensive sampling.
Measure: Median (Full Range); unit: hours
Arm/Group | REPLAGAL
Number analyzed (Participants) | 10
hours
  Week 0 | 40.000 [20.00 to 40.00]
  Week 28 | 40.000 [20.00 to 41.00]

25. Secondary Outcome: Volume of Distribution at Steady State (Vss) of REPLAGAL
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. V(ss) = (dose/AUC)*MRT, where MRT is mean residence time.
Time Frame: as for outcome 18
Population: Intensive PK Set included participants in the PK Set who provided intensive sampling.
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | REPLAGAL
Number analyzed (Participants) | 10
milliliters (mL)
  Week 0 | 7834 (1625.9)
  Week 28 | 12310 (16988)

26. Secondary Outcome: Volume of Distribution at Steady State Normalized Based on Body Weight of REPLAGAL
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Vss normalized for body weight was reported. V(ss) = [(dose/AUC)*MRT]/ body weight, where MRT is mean residence time.
Time Frame: as for outcome 18
Population: Intensive PK Set included participants in the PK Set who provided intensive sampling.
Measure: Mean (Standard Deviation); unit: milliliters per kilogram (mL/kg)
Arm/Group | REPLAGAL
Number analyzed (Participants) | 10
milliliters per kilogram (mL/kg)
  Week 0 | 135.9 (34.530)
  Week 28 | 202.1 (267.74)

27. Secondary Outcome: Dose Normalized Area Under Serum Concentration-time Curve From Time Zero to the Last Sampling Time (AUC0-last/Dose) of REPLAGAL
Description: AUC0-last/Dose was expressed using the unit: (minutes*units per milliliter)/(units per kilogram) [(min*U/mL)/(U/kg)].
Time Frame: as for outcome 18
Population: Intensive PK Set included participants in the PK Set who provided intensive sampling.
Measure: Mean (Standard Deviation); unit: (min*U/mL)/(U/kg)
Arm/Group | REPLAGAL
Number analyzed (Participants) | 10
(min*U/mL)/(U/kg)
  Week 0 | 0.005411 (0.0010847)
  Week 28 | 0.008119 (0.0044732)

28. Secondary Outcome: Dose Normalized Area Under the Serum Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-inf/Dose) of REPLAGAL
Time Frame: as for outcome 18
Population: Intensive PK Set included participants in the PK Set who provided intensive sampling.
Measure: Mean (Standard Deviation); unit: (min*U/mL)/(U/kg)
Arm/Group | REPLAGAL
Number analyzed (Participants) | 10
(min*U/mL)/(U/kg)
  Week 0 | 0.005520 (0.0010993)
  Week 28 | 0.008489 (0.0051204)

29. Secondary Outcome: Dose Normalized Maximum Observed Serum Concentration (Cmax/Dose) of REPLAGAL
Description: Cmax/Dose was expressed using the unit: (units/milliliter)/(units/kilogram) [(U/mL)/(U/kg)].
Time Frame: as for outcome 18
Population: Intensive PK Set included participants in the PK Set who provided intensive sampling.
Measure: Mean (Standard Deviation); unit: (U/mL)/(U/kg)
Arm/Group | REPLAGAL
Number analyzed (Participants) | 10
(U/mL)/(U/kg)
  Week 0 | 0.0001092 (0.000021579)
  Week 28 | 0.0001197 (0.000040471)

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to 14 days after EOT (up to Week 54)
Description: Safety Analysis Set included all participants in the ITT Set who received at least 1 dose of REPLAGAL.
Arm/Group | REPLAGAL
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | REPLAGAL (N=20)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Sepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | REPLAGAL (N=20)
Albuminuria (Renal and urinary disorders) | 2
Angina pectoris (Cardiac disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone metabolism disorder (Musculoskeletal and connective tissue disorders) | 2
COVID-19 (Infections and infestations) | 13
Chest discomfort (General disorders) | 2
Corneal opacity (Eye disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Haematuria (Renal and urinary disorders) | 2
Headache (Nervous system disorders) | 3
Oedema peripheral (General disorders) | 2
Pyrexia (General disorders) | 5
Upper respiratory tract infection (Infections and infestations) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT04974749/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT04974749/SAP_001.pdf